CLINICAL TRIAL: NCT02843152
Title: Risk Factor Analysis of Postoperative Cognitive Dysfunction and Its Association With Inflammation Related Gene Polymorphism
Brief Title: Association Study Postoperative Cognitive Dysfunction Associated With Inflammation Polymorphism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: dengji wang (Other)
Responsible Party: Sponsor-Investigator, dengji wang, Investigator, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Other Study IDs: 14038789
Record Dates: First submitted 2016-06-25; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: POCD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This study use Loewenstein cognitive function rating scale to meet the standards of the elderly cognitive function assessment. POCD diagnostic criteria used is the recommended value Z current international law, in order to reduce the effects of exercise, we selected 50 cases of patients with age-matched healthy control group as a spouse, the same scale testing. And Loewenstein Assessment Scale cognitive function after some domestic research proved to have good sensitivity, and easy to test small changes in cognitive ability.

Before the investigation began strict inclusion and exclusion criteria, the use of simple intelligence scale exclude preoperative cognitive decline in the elderly significantly, the use of depression rating scale for anxiety rating scale before surgery to exclude severe depression and severe anxiety in elderly self self patient. Testing by the same person in the same way neurocognitive assessment test twice, 7 days apart.

Studies in Chinese population, susceptibility SNPs and genetic POCD but there are few reports of this project uses 1: 1 matched case-control study, by comparison POCD SNPs and control groups of different polymorphisms, polymorphisms Discussion Han population of postoperative cognitive dysfunction associated with susceptibility to find Chinese Han population of postoperative cognitive disorders genetic susceptibility markers, which provide scientific screening and early diagnosis of postoperative cognitive impairment at high risk in accordance with

DETAILED DESCRIPTION:
1. study 1.1 The study inclusion criteria: The study in January 2015 - June 2015 Xuzhou Medical College Hospital orthopedic ward in elderly patients, level of education for primary ((0 <schooling ≤6). Check all other indicators of the patients were in the normal range, no liver, kidney, lung, heart and other organ dysfunction, the operation time was 60 ~ 180min, ASA classified as class II.

   1.2 study exclusion criteria: Severe vision (1) no history of cerebrovascular disease (2) Other medical history (3) No alcohol dependence and other substance abuse history (4) to cause central nervous system damage did not affect cognitive function can not affect cognitive tests, hearing and limb movement disorder (5) without mental illness (6) Exclude known preoperative cognitive dysfunction (7) can not articulate the patient's own meaning or do not match, the patient can not communicate very well.

   In contrast to cases by sex and age and frequency matching. Study subjects were Chinese Han population, and signed informed consent form, a collection of peripheral blood specimens (5mlEDTA anticoagulated blood). At the same time, by specially trained investigators to complete the epidemiological survey.
2. field epidemiology survey methodology 2.1 Questionnaire items (perioperative observations Indicator) 2.1.1 Preoperative: gender, age, education, past medical history (hypertension, diabetes, chronic lung disease), surgery.

2.1.2 Surgery: The operation time, the number of anesthesia, fentanyl, remifentanil, the dosage of atropine, hypotension, hypertension. Intraoperative hypotension cases: surgery or any time SBP≤90 mm Hg compared with preoperative blood pressure reduced by more than 30% for longer than 5min; intraoperative hypertension cases: surgery any time SBP≥140 / 90mmHg or comparing preoperative more than 30% increase in blood pressure over the duration of 5min.

2.1.3 Postoperative: Postoperative 7d or prior to discharge using a visual analog scale (vasual analogue scale, VAS) to assess the degree of pain the patient and postoperative complications were recorded (with or without infection, reoperation).

2.2 neuropsychological assessment tools: 2.2.1 Simple Intelligence Scale (Mini-Mental State Examination, MMSE) 2.2.2 Self-Rating Depression Scale (Self-Rating Depression Scale, SDS) 2.2.3 Self-Rating Anxiety Scale (Self-Rating Anxiety Scale SAS) 2.3.4 know Abilities Screening Instrument 2.3 postoperative cognitive dysfunction assessment program and criteria: POCD for assessment, the project recommended using the current Z value of international law, in order to reduce the effects of exercise, selected 50 cases of patients with age-matched healthy control group as a spouse, the same scale test, the exclusion criteria with the control group. POCD is calculated as: Z = (X-X reference) / SD .. X is a preoperative patient surgery, the score of the difference, X reference is the difference between the scale scores before and after the control group, SD is the standard deviation of the difference between the control group. When the Z value of the test in two or more scale test is greater than 1.96 is considered POCD.

Answers were recorded accurately complete the test score or the time required. MMSE scale is mainly used for screening in elderly subjects, excluding preoperative cognitive function in patients with significantly decreased. Self-Rating Depression Scale suitable for different age, gender patients with depression score. Self-Rating Anxiety Scale suitable for different age, gender patients' anxiety before surgery to evaluate anxiety and depression status, excluding severe anxiety and depression survey, no longer be evaluated cognitive abilities.

In addition, we selected 50 cases of patients with age-matched healthy control group as a spouse, learn to reduce the effects of neuropsychological tests before the subject later. Testing by the same person in the same way neurocognitive assessments, test twice, 7 days apart. Loewenstein cognitive function using standard rating scale for the assessment of cognitive function in older people. Loewenstein cognitive neuropsychological rating scale is Luria and Piaget's developmental model is based, including the time and place orientation, visual perception, spatial perception, action apply, depending on the sports organization, logical thinking, attention and concentration, assessment the project was more than MMSE, and a detailed breakdown can not only reflect the patient's cognitive problems in these areas, but also to predict the progress of change and prognosis of brain injury, a more appropriate amount is used to assess postoperative cognitive impairment table.

In this study, an international research organization POCD recommended Z-score method to determine the incidence of postoperative cognitive dysfunction, and is divided into POCD and control groups. To analyze the effect of learning, healthy control subjects before and after the calculation of each individual test item score difference, the difference between the results of mean and standard deviation, and then calculated for each patient before and after surgery score difference between the individual test items, use When this difference is divided by the standard deviation that is obtained by subtracting the mean of each individual test item Z-score, Z score greater the greater the decline after the test scores compared with preoperative. Each individual test items Z summing points, healthy control subjects Z points and calculate the standard deviation S, each patient divided by the S and Z-score is the composite of the patient's Z-score, if the composite Z-score ≥21.96 individual tests or have two or more Z-score greater than or equal 96, it is considered that the patients POCD. Orthopedic patients in the control group from the same period, the age and gender of the patient group want to match.

2.4 survey items related definitions 2.4.1 alcohol. Drinking 2 years and above, equivalent to an ethanol content of women ≥20 g / d, male ≥40 g / d.

2.4.2 Hypertension. Are receiving antihypertensive medications, or past medical history of diagnosed hypertension, or in patients with more than 2 times extraordinary Systolic ≥140 mmH; and (or) DBP) 90 mmHg} 2.4.3 diabetes. Taking hypoglycemic drugs, or a previous diagnosis of diabetes or fasting glucose measurement ≥7.0 mmol / L, random blood glucose ≥11.1 mmol / L.

2.4.4 TNM staging. Use appropriate staging of the disease 2.4.5 intraoperative hypotension. A reduction in blood pressure than before anesthesia or 20% less than 80 mmHg systolic 2.4.6 postoperative continuous analgesia. Surgery received intravenous analgesia pump, intravenous analgesia with fentanyl as postoperative analgesics, loading dose of 0.5μg / kg, background dosage 0. 3μg / (kg • h), a single dose of 0.25μg / kg , lockout time 15 min, time 48 h.

ELIGIBILITY:
Inclusion Criteria:

* Education for primary ((0 <schooling ≤6)
* The operation time was 60 ~ 180min
* ASA classification as Class II

Exclusion Criteria:

* No history of cerebrovascular disease
* No history of central nervous system injury caused by the impact of other cognitive functions
* No alcohol dependence and other substance abuse history
* No vision can severely affect cognitive tests, hearing and limb movement disorder

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects were Chinese Han population,Xuzhou Medical College Hospital orthopedic ward in elderly patients
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Determine the relevance of inflammation-related genes and SNPs of susceptible POCD | 1 year
  In this study of an international research organization POCD recommended Z-score method to determine postoperative cognitive dysfunction, and is divided into POCD and non POCD group, if the composite Z-score ≥1.96 or have two or more individual test Z-score greater than or equal 1.96 considers the patient POCD group, otherwise non POCD group. They were recorded POCD group and non-POCD group education of patients, medical history, surgery time, anesthesia time, and the amount of narcotic drugs, hypotension, hypertension, postoperative pain, complications, smoking, drinking, blood samples were analyzed patient patients with IL-1β, IL-6, IL-10, VDR, BDNF gene polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: junli cao, Study Chair — Jiangsu Key Laboratory of Anesthesiology chinese
Locations (1):
- Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided